CLINICAL TRIAL: NCT00633945
Title: Evaluation of Lenalidomide (REVLIMID®) in Cutaneous LE: A Prospective, Non Controlled, Open Label Pilot Study to Evaluate the Off-Label Use of the FDA-approved Drug Lenalidomide (REVLIMID®) in Patients With Cutaneous Lupus Erythematosus
Brief Title: Evaluation of Lenalidomide (REVLIMID®) to Treat Subjects With Cutaneous Lupus Erythematosus (CLE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 806259
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Cutaneous Lupus Erythematosus (CLE)
Keywords: Cutaneous Lupus Erythematosus; CLE; lenalidomide; revlimid; thalidomide derivative; drug; lupus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): Open label lenalidomide received.
  Interventions: Drug: Lenalidomide
- Lenalidomide 2 (Experimental): Open label lenalidomide received.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of lenalidomide (Revlimid®) in subjects with Cutaneous Lupus Erythematosus (CLE). The study drug will be used in an off-label indication to treat 6 subjects for 12 months each. Men and women over the age of 18, who have a biopsy proven diagnosis of CLE and who have failed standard treatment, will be included in the study.

DETAILED DESCRIPTION:
Cutaneous lupus erythematosus (CLE) is a chronic and often disabling disease which affects the skin. Many patients experience scarring and inflammation of the skin, which often occur on the face. Moderate to severe CLE is most frequently treated with antimalarial drugs such as hydroxychloroquine, quinacrine or chloroquine. Up to 70% of CLE patients treated with antimalarials experience a beneficial clinical response, while the remainder of patients show no response or continue to experience progression of the disease. Thalidomide has been used successfully in such patients, with up to 75% clinical response rate in refractory CLE patients. However, thalidomide is a known teratogen and can cause severe birth defects, including short, malformed limbs and damage to peripheral nerves in the extremities, requiring patients to be monitored for pregnancy. In addition, up to 25% of patients on thalidomide develop peripheral neuropathy. A new drug, lenalidomide (REVLIMID®), an analogue of thalidomide, has been developed to treat neoplastic and inflammatory conditions, including various oncologic conditions such as multiple myeloma, myelodysplastic syndrome and solid tumors. Unlike thalidomide, lenalidomide (REVLIMID®) is not known to cause the extent of serious side effects caused by thalidomide; however, it must also be monitored for side effects and be distributed under the RevAssist program authorized by the drug manufacturer, Celgene Corporation.

The primary goal of this investigator-initiated, small pilot study is to evaluate the safety and effectiveness of lenalidomide (REVLIMID®) in CLE subjects using measurements such as the CLASI (Cutaneous Lupus Activity and Severity Index). The study drug will be used in an off-label indication to treat 6 subjects, for whom lenalidomide (REVLIMID®) will be provided at no cost by the drug manufacturer. Men and women over the age of 18, who have a biopsy proven diagnosis of refractory CLE and who have failed standard treatment with hydroxychloroquine for up to three months, will be included in the study. Secondarily, the study will evaluate the biologic effects of lenalidomide on pathogenic and immunologic mechanisms of the CLE disease process during the treatment period by collecting skin specimens (biopsies) and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must understand and voluntarily sign Informed Consent and HIPAA forms.
* Males and females over the age of 18 at the time of signing informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements
* Subjects must have biopsy proven Cutaneous Lupus Erythematosus (CLE) either in the form of Discoid Lupus Erythematosus (DLE) or Subacute Lupus Erythematosus (SCLE), with or without systemic involvement.
* Subjects must have grade II erythema in at least three skin locations as defined by the Cutaneous Lupus Activity and Severity Index (CLASI).
* Subjects must have failed standard treatment with hydroxychloroquine (Plaquenil) for up to three months.
* Female subjects who are not pregnant.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional method AT THE SAME TIME, at least 28 days before starting to take lenalidomide (Revlimid®). FCBP must also agree to ongoing pregnancy testing. Males must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* If pregnancy or a positive pregnancy test is noted in a study subject or in the partner of a male study subject during study participation, the study drug must be discontinued immediately.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality or psychiatric illness that would prevent the subject from signing the informed consent form.
* Female subjects who are pregnant, plan to be pregnant during the study, or who are breastfeeding.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk for study participation, or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Prior history of deep vein thrombosis (DVT).
* Prior history of pulmonary embolus (PE).
* Known positive for HIV viral DNA by qPCR.
* Positive hepatitis B surface antigen, or hepatitis C.
* Platelet count < 50,000/mcL.
* Absolute neutrophil count < 750/mcL
* Lymphopenia < 500/mcL.
* Have current signs or symptoms of severe progressive or uncontrolled renal disease (creatinine ≥1.5 x ULN).
* If female, unwillingness to use one highly effective method and one additional method of birth control.
* If male, unwillingness to use a latex condom during intercourse with females of childbearing potential.
* Continued therapy with thalidomide.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-11; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria P Werth, MD, Principal Investigator — University of Pennsylvania, Department of Dermatology
Locations (1):
- Hospital of the University of Pennsylvania, Department of Dermatology, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Okon L, Rosenbach M, Krathen M, Rose M, Propert K, Okawa J, Werth V. Lenalidomide in treatment-refractory cutaneous lupus erythematosus: Efficacy and safety in a 52-week trial. J Am Acad Dermatol. 2014 Mar;70(3):583-4. doi: 10.1016/j.jaad.2013.11.007. No abstract available. PMID 24528907

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The sample size was determined by the number of study subjects for whom Celgene Corporation was willing to supply medication during and beyond the study period. It was felt that 5 study subjects would provide valuable information about the responsiveness of severe CLE to lenalidomide (REVLIMID®) and subjects' tolerability to the study medication.
Groups:
- Lenalidomide: Patients took 5 mg daily of oral lenalidomide for the initial 6 weeks. Patients who had responded at 6 weeks lowered their dose to 5 mg every other day, while non-responders were increased to a dose of 10 mg daily.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 5
Completed | 3
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (4.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Lupus Area and Severity Index (CLASI)
Description: The Cutaneous Lupus Area and Severity Index (CLASI); range of disease activity is 0-70. Lower scores reflect less activity.
Time Frame: Weeks 0 through 52
Population: Two patients were not included at week 52 because one did not respond and one had new onset proteinuria and arthralgias.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  0 weeks | 21.4 [16 to 26]
  6 weeks | 10.8 [8 to 18]
  12 weeks | 8.6 [1 to 18]
  52 weeks: number analyzed (Participants) | 3
  52 weeks | 5.3 [0 to 12]

2. Secondary Outcome: Number of Participants With Change in IFN and CD4 Levels at 6 Weeks
Description: CXCL10, an interferon-inducible chemokine, and immunophenotyping by immunostaining. Measurement of interferon-inducible genes from peripheral blood mononuclear cells before and after treatment.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Lenalidomide Responders: Response with CLASI
- Lenalidomide Nonresponder: Lack of response with CLASI
Arm/Group | Lenalidomide Responders | Lenalidomide Nonresponder
Number analyzed (Participants) | 4 | 1
Participants
  IFN score decrease | 4 | 1
  CD4 decrease | 4 | 1

3. Secondary Outcome: Physician Global Assessment (PGA) for Skin
Description: General skin scores were recorded on a 10 cm visual analogue scale at each visit. At each visit on scale 0-10, 0 corresponding to worst skin condition imaginable and 10 to perfect health.
Time Frame: Weeks 0 through 52
Population: 5 patients until week 12, 3 patients to week 52. Dropout prevented proper analysis of week 12 to 52.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  week 0 | 6 [0 to 10]
  week 6 | 3 [0 to 10]
  week 12 | 3.8 [0 to 10]
  week 52: number analyzed (Participants) | 3
  week 52 | 2 [0 to 10]

4. Secondary Outcome: Patient General Assessment (PtGA) for Skin
Description: General skin scores were recorded by the patient on a 10 cm visual analogue scale at each visit by the patient. At each visit on scale 0-10, 0 corresponding to worst skin condition imaginable and 10 to perfect health.
Time Frame: Weeks 0 through 52
Population: 5 patients until week 12, 3 patients to week 52. Dropout prevented proper analysis of week 12 to 52.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  week 0 | 5.6 [0 to 10]
  week 6 | 3.6 [0 to 10]
  week 12 | 4.2 [0 to 10]
  week 52: number analyzed (Participants) | 3
  week 52 | 0.8 [0 to 10]

5. Secondary Outcome: Pain in Skin
Description: Pain in skin was recorded on a 10 cm visual analogue scale at each visit by the patient. At each visit on scale 0-10, 0 corresponding to no pain and 10 to pain as bad as you can imagine.
Time Frame: Weeks 0 through 52
Population: 5 patients until week 12, 3 patients to week 52. Dropout prevented proper analysis of week 12 to 52.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  week 0 | 4.5 [0 to 10]
  week 6 | 2 [0 to 10]
  week 12 | 2.5 [0 to 10]
  week 52: number analyzed (Participants) | 3
  week 52 | 0.5 [0 to 10]

6. Secondary Outcome: Itch in Skin
Description: Itch scores were recorded on a 10 cm visual analogue scale at each visit by the patient. At each visit on scale 0-10, 0 corresponding to no itch and 10 to itch as bad as you can imagine.
Time Frame: Weeks 0 through 52
Population: 5 patients until week 12, 3 patients to week 52. Dropout prevented proper analysis of week 12 to 52.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  week 0 | 4.0 [0 to 10]
  week 6 | 1.2 [0 to 10]
  week 12 | 2.25 [0 to 10]
  week 52: number analyzed (Participants) | 3
  week 52 | 0 [0 to 10]

7. Secondary Outcome: Fatigue
Description: Fatigue scores were recorded on a 10 cm visual analogue scale at each visit by the patient. At each visit on scale 0-10, 0 corresponding to no fatigure and 10 to fatigue as bad as you can imagine.
Time Frame: Weeks 0 through 52
Population: 5 patients until week 12, 3 patients to week 52. Dropout prevented proper analysis of week 12 to 52.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  week 0 | 7.25 [0 to 10]
  week 6 | 3.4 [0 to 10]
  week 12 | 5.25 [0 to 10]
  week 52: number analyzed (Participants) | 3
  week 52 | 3 [0 to 10]

8. Secondary Outcome: Skindex Symptoms
Description: Skindex symptoms scores are scored 1-5 and then normalized to 100, with a higher score corresponding to a worse impression. The absence of symptom impact on QoL is scored as "20" (this is represented as a 1 on the 1-5 scale. The worst impact of symptoms on QoL is 100. This is represented as a 5 on the 1-5 scale.
Time Frame: Weeks 0 through 52
Population: 5 patients until week 12, 3 patients to week 52. Dropout prevented proper analysis of week 12 to 52.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  week 0 | 58.5 [0 to 100]
  week 6 | 41.82 [0 to 100]
  week 12 | 36.4 [0 to 100]
  week 52: number analyzed (Participants) | 3
  week 52 | 12.5 [0 to 100]

9. Secondary Outcome: Skindex Function
Description: Skindex function scores are scored 1-5 and then normalized to 100, with a higher score corresponding to a worse impression. The absence of function impact on QoL is scored as "20" (this is represented as a 1 on the 1-5 scale. The worst impact of function on QoL is 100. This is represented as a 5 on the 1-5 scale.
Time Frame: Weeks 0 through 52
Population: 5 patients until week 12, 3 patients to week 52. Dropout prevented proper analysis of week 12 to 52.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Lenalidomide
Number analyzed (Participants) | 5
units on a scale
  week 0 | 41.26 [0 to 100]
  week 6 | 30.42 [0 to 100]
  week 12 | 29.2 [0 to 100]
  week 52: number analyzed (Participants) | 3
  week 52 | 4.2 [0 to 100]

ADVERSE EVENTS:
Groups:
- Group 1: Lenalidomide treated patients
Arm/Group | Group 1
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
This study is limited by small sample size and open label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No